CLINICAL TRIAL: NCT02810379
Title: Combination of Video and Written Information Provides the Patient With a More Comprehensive Level of Knowledge About Endoscopic Retrograde Cholangiopancreatography: Study Protocol for Randomized Controlled Trial
Brief Title: Video Consent Form Versus Written Consent Form for ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ERCP-1
Record Dates: First submitted 2016-04-25; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Consent Forms of ERCP
Keywords: informed consent; ERCP; video

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- written informed consent (Placebo Comparator): participants read the written informed consent documents befor ERCP
  Interventions: Procedure: written informed consent
- video+written informed consent (Experimental): participants watch a video about the ERCP and read the written informed consent documents before ERCP
  Interventions: Procedure: video+written informed consent

INTERVENTIONS:
Procedure: written informed consent
  Arms: written informed consent
Procedure: video+written informed consent
  Arms: video+written informed consent

SUMMARY:
To prove that video about endoscopic retrograde cholangiopancreatography (ERCP) combined with written informed consent provides participants more information about the procedure, which can make participants understand the procedure well. Investigators advocate the development of institutional and national guidelines to ensure optimal practices of acquiring informed consent.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients who will receive ERCP

Exclusion Criteria:

* under 18 years or more than 70 years
* pregnancy or breast-feeding women
* circulatory and respiratory disorders
* mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
time for informed consent practices before ERCP | 2 days
time for extra explanation about ERCP | 2 days

SECONDARY OUTCOMES:
satisfaction degree about the informed consent practices | 2 days

OTHER OUTCOMES:
anxiety level after the informed consent practices | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

REFERENCES:
- [Derived] Xia T, Zhu YB, Zeng YB, Chen C, Wang SL, Zhao SB, Su XJ, Wang D, Yao J, Li ZS, Bai Y. Video education can improve awareness of risks for patients undergoing endoscopic retrograde cholangiopancreatography: A randomized trial. J Dig Dis. 2019 Dec;20(12):656-662. doi: 10.1111/1751-2980.12824. Epub 2019 Nov 21. PMID 31618520